CLINICAL TRIAL: NCT02756819
Title: International Multicentre, Observational, Non-Interventional Prospective Study of Azilsartan Medoxomil in Patients With Arterial Hypertension Who Are Overweight or Obese in the Russian Federation and The Republic of Kazakhstan
Brief Title: International Multicenter, Observational, Non-Interventional Prospective Study of Azilsartan Medoxomil in Participants With Arterial Hypertension Who Are Overweight or Obese in the Russian Federation and The Republic of Kazakhstan
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Azilsmedox-5008; MACS-2014-100663 (Other: Takeda)
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azilsartan Medoxomil: Overweight or obese participants with hypertension who received azilsartan medoxomil tablets, orally, as prescribed by physician according to local summary of product characteristics (SmPC) were observed for approximately 6 months.
  Interventions: Drug: Azilsartan Medoxomil

INTERVENTIONS:
Drug: Azilsartan Medoxomil — Azilsartan medoxomil tablets
  Other Names: Edarbi®

SUMMARY:
The purpose of this study is to estimate antihypertensive effect of azilsartan medoxomil (Edarbi®) therapy on blood pressure in participants with overweight or obesity in routine clinical practice of hypertension (HTN) treatment in the Russian Federation and in the Republic of Kazakhstan..

DETAILED DESCRIPTION:
The drug being tested in this study is called azilsartan medoxomil (Edarbi®). Azilsartan medoxomil is being tested to treat people who have hypertension. This study looks at the clinic systolic and diastolic blood pressure (SBP, DBP) in obese participants who were prescribed azilsartan medoxomil by physicians.

The study enrolled 1945 patients. All participants were asked to take azilsartan medoxomil as prescribed by their physician according to local SmPC.

This multi-center trial was conducted in the Russian Federation and the Republic of Kazakhstan. The overall duration of study for observation was approximately 6 months. Participants made multiple visits to the clinics as assigned by each physician according to their routine practice, in every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age with hypertension 1-2 grade.
2. Participants with:

   * newly diagnosed arterial HTN or
   * inadequately controlled previously prescribed monotherapy with Renin-Angiotensin-Aldosterone System (RAAS) blocker or
   * inadequately controlled previously prescribed combination therapy with RAAS blocker + diuretic or RAAS blocker + calcium antagonist.
3. The physician decides to prescribe Edarbi®

   * as monotherapy or
   * as a part of combination therapy including diuretics or calcium antagonists;
4. Overweight or obesity of any degree (body mass index> 25 kg/m^2);
5. Is capable of understanding the written informed consent, provides signed and written informed consent, and agrees to comply with protocol requirements. In case the participant is blind or unable to read, informed consent will also be witnessed.

Exclusion Criteria:

1. Confirmed secondary HTN;
2. Contraindications for Edarbi® of respective approved local summary of product characteristics (SmPC) of Edarbi®;
3. Any reasons of medical and non-medical character, which in the opinion of the physician can prevent participant participation in the study.
4. Is an employee or family member of the investigator or study site personnel.
5. Is currently participating in a clinical trial. Participation in non-interventional registries is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight or obese participants with Hypertension (HTN) grade 1-2 were observed.
Sampling Method: Non-Probability Sample
Enrollment: 1945 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (65):
- Kazakhstan (7):
  - JSC Central Clinical hospital, Almaty
  - Research Institute of Cardiology and Internal Diseases, Almaty
  - Kazakh Medical University of Continuing Education, Almaty
  - Central Clinical Hospital, Almaty
  - National Scientific center of oncology and transpontology, Astana
  - Karaganda State Medical Academy, Karaganda
  - Semipalatinsk State Medical Academy, Semey
- Russia (58):
  - Altay regional cardiological center, Barnaul
  - Belgorod Regional Clinical Hospital of St. Joasaph, Belgorod
  - Bryansk Regional Cardiological center, Bryansk
  - Medical center Lotos, Chelyabinsk
  - Regional clinical Hospital #3, Chelyabinsk
  - Istochnik Clinic, Chelyabinsk
  - Medical Center Academy of Health, Chita
  - Chita State Medical Academy, Chita
  - Regional Clinical Consultative Diagnostic center, Irkutsk
  - Cardiological center, Ivanovo
  - Consultative Diagnostic Center Ministry of Health of Udmurt Republic, Izhevsk
  - City clinical hospital #2 sosnovaya roscha, Kaluga
  - Kemerovo Regional Clinical Cardiological center named after Barabash L.S., Kemerovo
  - Kemerovo Regional Clinical hospital named after Belyaev S.V., Kemerovo
  - Regional Clinical Hospital #1 named after S.I.Sergeev, Khabarovsk
  - Road clinical hospital at the station Khabarovsk JSC "Russian Railways", Khabarovsk
  - Northern Clinical Emergency Hospital, Kirov
  - Kirov Clinical hospital named after Yurlova V.I., Kirov
  - Kostroma Regional Clinical Hospital named after Korolev E.I., Kostroma
  - Lipetsk City policlinic #7, Lipetsk
  - LLC Medical center Semeynyiy doctor, Magnitogorsk
  - City policlinic #166, branch 1, Moscow
  - City policlinic #166, branch 2, Moscow
  - City clinical hospital #1 named after N.I. Pirogova, Moscow
  - City polyclinic #22, Moscow
  - City polyclinic #11,branch #1, Moscow
  - City polyclinic #11, Moscow
  - City polyclinic #11, branch #3, Moscow
  - Volga District Medical Centre (VDMC) under Federal Medical and Biological Agency (FMBA), Nizhny Novgorod
  - Omsk state medical university, Omsk
  - Medical Center "Novaya medicina", Orekhovo-Zuyevo
  - Penza Regional Clinical hospital named after N.N. Burdenko, Penza
  - Regional clinical hospital named after N.N. Burdenko, Penza
  - Clinical Cardiological Center, Perm
  - Road Clinical Hospital at the Rostov-Ch. JSC Russian Railways, Rostov-on-Don
  - Rostov State Medical University, Rostov-on-Don
  - City Consultative Diagnostic Center #1, Saint Petersburg
  - City polyclinic #117, Saint Petersburg
  - CJSC Cardioclinic, Saint Petersburg
  - City Consultative Diagnostic Clinic#1 Primorsky District, Diabetological center #5, Saint Petersburg
  - City polyclinic #14, Samara
  - Samara Regional Clinical Cardiological center, Samara
  - Saratov city polyclinic #2, Saratov
  - LLC Multiprofile medical clinic Sova, Saratov
  - City polyclinic #3, Tomsk
  - Scientific Research Institute of Cardiology, Tomsk
  - Tomsk Clinical hospital, Tomsk
  - Regional Clinical Cardiological center, Tver'
  - Tyumen Cardiological center, Tyumen
  - Regional Cardiological center, Ulyanovsk
  - City hospital #4, Vladimir
  - Volgograd Regional Clinical hospital #1, Volgograd
  - Volgograd Regional Clinical Cardiological center #1, Volgograd
  - Voronezh Regional Clinical Diagnostic center, Voronezh
  - Voronezh City Clinical polyclinic #4, Voronezh
  - National Medical Center, Yakutsk
  - Yaroslavl Regional Clinical Hospital of War Veterans, Yaroslavl
  - Medical AssociationNew Hospital, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 65 sites in the study in Russian Federation and the Republic of Kazakhstan from 18-Jul-2016 to 08-May-2018.
Pre-assignment Details: Participants with a diagnosis of hypertension and who were obese, prescribed azilsartan medoxomil in accordance with local summary of product characteristics (SmPC) were enrolled in this observational study.
Groups:
- Azilsartan Medoxomil: Overweight or obese participants with hypertension who received azilsartan medoxomil tablets, orally, as prescribed by physician according to local SmPC were observed for approximately 6 months.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil
Started | 1945
Per-protocol Set (PPS) | 1724 (Participants who were enrolled, received Edarbi® therapy and did not have major protocol deviations.)
Safety Analysis Set (SAS) | 1934 (Participants who received at least one dose of Edarbi® therapy and had any follow-up data.)
Completed | 1893
Not Completed | 52
Not completed — Lost for observation | 23
Not completed — Patient's unwillingness | 16
Not completed — Insufficient efficacy | 2
Not completed — Adverse Event | 2
Not completed — Reason not Specified | 9

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received azilsartan medoxomil.
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed is the number of participants with data available for analysis at the given timepoint.
  years
    number analyzed (Participants) | 1944
    (all) | 55.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1103
  Male | 842
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European | 1787
  Asian | 158
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 1759
  Kazakhstan | 186

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Systolic Blood Pressure (SBP) at Month 6
Description: The change in clinic sitting SBP measured at Month 6 relative to baseline.
Time Frame: Baseline and Month 6
Population: Full analysis set (FAS) included all participants who were enrolled and received azilsartan medoxomil (Edarbi®) therapy. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
mmHg
  Baseline | 156.8 (11.8)
  Change from baseline at Month 6: number analyzed (Participants) | 1890
  Change from baseline at Month 6 | -30.5 (13.4)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change at Month 6 relative to Baseline

2. Secondary Outcome: Change From Baseline in Clinic Diastolic Blood Pressure (DBP) at Month 6
Description: The change in clinic sitting DBP measured at Month 6 relative to baseline.
Time Frame: Baseline and Month 6
Population: FAS included all participants who were enrolled and received azilsartan medoxomil (Edarbi®) therapy. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
mmHg | -14 (9.4)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change at Month 6 relative to Baseline

3. Secondary Outcome: Percentage of Participants With Response at Month 6
Description: Response was defined as a decrease of SBP ≥20 mm Hg or a decrease of DBP ≥10 mm Hg.
Time Frame: Month 6
Population: Participants from FAS, all participants who were enrolled and received azilsartan medoxomil (Edarbi®) therapy with data available for analysis at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1890
percentage of participants | 92.6 [91.3 to 93.7]

4. Secondary Outcome: Percentage of Participants Who Achieved Target Blood Pressure (BP) SBP<140 mm Hg and DBP<90 mm Hg
Time Frame: Month 6
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1890
percentage of participants | 86.4 [84.8 to 87.9]

5. Secondary Outcome: Change From Baseline in Clinic Systolic Blood Pressure (SBP) in Subgroups of Participants at Month 6
Description: The change in clinic sitting SBP measured at Month 6 relative to baseline. Subgroups included overweight, obesity I (basic metabolic rate [BMI] 30-34.9), class II (BMI 35-39.9) and class III (BMI ≥ 40), impaired glucose tolerance, normal glucose metabolism, diabetes mellitus (Yes/No), metabolic syndrome, neither diabetes mellitus (DM) nor metabolic syndrome.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
mmHg
  Change at Week 6, Overweight: number analyzed (Participants) | 616
  Change at Week 6, Overweight | -30.2 (13.6)
  Change at Week 6, BMI (Obesity class I): number analyzed (Participants) | 860
  Change at Week 6, BMI (Obesity class I) | -30.6 (13.2)
  Change at Week 6, BMI (Obesity class II): number analyzed (Participants) | 320
  Change at Week 6, BMI (Obesity class II) | -31.5 (12.5)
  Change at Week 6, BMI (Obesity class III): number analyzed (Participants) | 93
  Change at Week 6, BMI (Obesity class III) | -27.1 (15.8)
  Change at Week 6, Normal glucose metabolism: number analyzed (Participants) | 1455
  Change at Week 6, Normal glucose metabolism | -30.5 (13.3)
  Change at Week 6, Impaired glucose tolerance: number analyzed (Participants) | 205
  Change at Week 6, Impaired glucose tolerance | -30.1 (13.2)
  Change at Week 6, Diabetes Mellitus (No): number analyzed (Participants) | 1467
  Change at Week 6, Diabetes Mellitus (No) | -30.6 (13.3)
  Change at Week 6, Diabetes Mellitus (Yes): number analyzed (Participants) | 230
  Change at Week 6, Diabetes Mellitus (Yes) | -30.5 (13.7)
  Change at Week 6,Neither DM nor Metabolic Syndrome: number analyzed (Participants) | 698
  Change at Week 6,Neither DM nor Metabolic Syndrome | -29.4 (13.6)
  Change at Week 6, Metabolic syndrome: number analyzed (Participants) | 962
  Change at Week 6, Metabolic syndrome | -31.2 (13.1)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Overweight)
Statistical Analysis 2: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class I)
Statistical Analysis 3: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class II)
Statistical Analysis 4: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class III)
Statistical Analysis 5: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test; P-value was reported for Change from baseline at Month 6 (Normal glucose metabolism)
Statistical Analysis 6: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Impaired glucose tolerance)
Statistical Analysis 7: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Diabetes Mellitus - No)
Statistical Analysis 8: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Diabetes Mellitus - Yes)
Statistical Analysis 9: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Neither diabetes mellitus nor metabolic syndrome)
Statistical Analysis 10: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Metabolic syndrome)

6. Secondary Outcome: Change From Baseline in Clinic Diastolic Blood Pressure (DBP) in Subgroups of Participants at Month 6
Description: The change in clinic sitting DBP measured at Month 6 relative to baseline. Subgroups included overweight, obesity I (basic metabolic rate [BMI] 30-34.9), class II (BMI 35-39.9) and class III (BMI ≥ 40), impaired glucose tolerance, normal glucose metabolism, diabetes mellitus (Yes/No), metabolic syndrome, neither diabetes mellitus nor metabolic syndrome.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
percentage of participants
  Change at Week 6, Overweight: number analyzed (Participants) | 616
  Change at Week 6, Overweight | -13.9 (9.5)
  Change at Week 6, BMI (Obesity class I): number analyzed (Participants) | 860
  Change at Week 6, BMI (Obesity class I) | -14 (9.3)
  Change at Week 6, BMI (Obesity class II): number analyzed (Participants) | 320
  Change at Week 6, BMI (Obesity class II) | -14.3 (9.4)
  Change at Week 6, BMI (Obesity class III): number analyzed (Participants) | 93
  Change at Week 6, BMI (Obesity class III) | -12.6 (11)
  Change at Week 6, Normal glucose metabolism: number analyzed (Participants) | 1455
  Change at Week 6, Normal glucose metabolism | -14 (9.4)
  Change at Week 6, Impaired glucose tolerance: number analyzed (Participants) | 205
  Change at Week 6, Impaired glucose tolerance | -14.2 (8.6)
  Change at Week 6, Diabetes Mellitus (No): number analyzed (Participants) | 1467
  Change at Week 6, Diabetes Mellitus (No) | -13.9 (9.2)
  Change at Week 6, Diabetes Mellitus (Yes): number analyzed (Participants) | 230
  Change at Week 6, Diabetes Mellitus (Yes) | -13.7 (10.6)
  Change at Week 6,Neither DM nor metabolic syndrome: number analyzed (Participants) | 698
  Change at Week 6,Neither DM nor metabolic syndrome | -13.4 (9.5)
  Change at Week 6, Metabolic syndrome: number analyzed (Participants) | 962
  Change at Week 6, Metabolic syndrome | -14.4 (9.1)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Overweight)
Statistical Analysis 2: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class I)
Statistical Analysis 3: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class II)
Statistical Analysis 4: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Obesity class III)
Statistical Analysis 5: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Normal glucose metabolism)
Statistical Analysis 6: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Impaired glucose tolerance)
Statistical Analysis 7: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Diabetes Mellitus - No)
Statistical Analysis 8: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Diabetes Mellitus - Yes)
Statistical Analysis 9: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Neither diabetes mellitus nor metabolic syndrome)
Statistical Analysis 10: Comparison: Azilsartan Medoxomil; Test type: Other; p < 0.001, Wilcoxon test — P-value was reported for Change from baseline at Month 6 (Metabolic syndrome)

7. Secondary Outcome: Percentage of Participants Who Achieved Target Blood Pressure (BP) in Subgroups of Participants at Month 6
Description: Target BP was SBP<140 mm Hg and DBP<90 mm Hg. Subgroups included BMI, overweight, Obesity I (BMI 30-34.9), class II (BMI 35-39.9) and class III (BMI ≥ 40), impaired glucose tolerance (Yes/No), metabolic syndrome (Yes/No) and diabetes mellitus (Yes/No).
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 1945
percentage of participants
  BMI (Overweight): number analyzed (Participants) | 553
  BMI (Overweight) | 89.8 [87.1 to 92.1]
  BMI (Obesity Class I): number analyzed (Participants) | 746
  BMI (Obesity Class I) | 86.7 [84.3 to 88.9]
  BMI (Obesity Class II): number analyzed (Participants) | 264
  BMI (Obesity Class II) | 82.5 [77.9 to 86.5]
  BMI (Obesity Class III): number analyzed (Participants) | 69
  BMI (Obesity Class III) | 74.2 [64.1 to 82.7]
  Normal glucose metabolism: number analyzed (Participants) | 1280
  Normal glucose metabolism | 88 [86.2 to 89.6]
  Impaired glucose tolerance: number analyzed (Participants) | 165
  Impaired glucose tolerance | 80.5 [74.4 to 85.7]
  Diabetes Mellitus (No): number analyzed (Participants) | 1268
  Diabetes Mellitus (No) | 86.4 [84.6 to 88.1]
  Diabetes Mellitus (Yes): number analyzed (Participants) | 188
  Diabetes Mellitus (Yes) | 81.7 [76.1 to 86.5]
  Neither diabetes mellitus nor metabolic syndrome: number analyzed (Participants) | 617
  Neither diabetes mellitus nor metabolic syndrome | 88.4 [85.8 to 90.7]
  Metabolic syndrome: number analyzed (Participants) | 828
  Metabolic syndrome | 86.1 [83.7 to 88.2]

ADVERSE EVENTS:
Time Frame: Baseline up to Month 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety population included all participants who received at least one dose of study treatment and had any follow-up data.
Arm/Group | Azilsartan Medoxomil
All-Cause Mortality (participants affected / at risk) | 0/1934
Serious Adverse Events (participants affected / at risk) | 6/1934
Other Adverse Events (participants affected / at risk) | 39/1934
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil (N=1934)
Angioedema (Skin and subcutaneous tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil (N=1934)
Hypotension (Vascular disorders) | 14
Hypertension (Vascular disorders) | 4
Dizziness (Nervous system disorders) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Left ventricular hypertrophy (Cardiac disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Palpitations (Cardiac disorders) | 1
Blood cholesterol increased (Investigations) | 1
Blood pressure decreased (Investigations) | 2
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Asthenia (General disorders) | 1
Headache (Nervous system disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Drug effect increased (General disorders) | 1
Drug ineffective (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT02756819/SAP_000.pdf
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02756819/Prot_001.pdf